CLINICAL TRIAL: NCT00213681
Title: CPAP Boussignac Versus Bilevel Pressure Support Ventilation in Severe Acute Cardiogenic Pulmonary Edema
Brief Title: CPAP Versus Bilevel Pressure Support Ventilation in Cardiogenic Pulmonary Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001/059/HP
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Severe Acute Cardiogenic Pulmonary Edema
Keywords: Pulmonary edema, respiratory failure, pressure support ventilation, continuous positive pressure
MeSH Terms: conditions — Pulmonary Edema; Respiratory Insufficiency

INTERVENTIONS:
Device: Boussignac CPAP - bilevel ventilation support

SUMMARY:
To evaluate whether bilevel positive airway pressure more rapidly improves ventilation than continuous positive airway pressure (CPAP) in patients with acute pulmonary edema. CPAP is delivered via a simple device connected to oxygen.

ELIGIBILITY:
Inclusion Criteria:

* age > 16 yrs, acute onset of severe respiratory distress, bilateral rales and typical findings of congestion on chest radiograph
* breathing frequency of > 30/min, SpO2 >90%, use of accessory respiratory muscles

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-11; Study Completion 2005-03

PRIMARY OUTCOMES:
Improvement in PaCO2 at the end of ventilation

SECONDARY OUTCOMES:
Endotracheal intubation, myocardial infarction and mortality during the first 24 hours
Duration of the ventilation
Blood gases, vital signs
Time to transfer to medical ward
Time to hospital discharge
Easiness to use was evaluated by nurses
Patients operational tolerance
Complications of each ventilation mode

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne MORITZ, MD, Principal Investigator — University Hospital, Rouen